CLINICAL TRIAL: NCT00050414
Title: Phase 2 Study of Efficacy and Safety of Trabectedin in Subjects With Advanced Ovarian Cancer
Brief Title: A Study of Trabectedin in Patients With Advanced Ovarian Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: PharmaMar (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR004057; ET743-INT-11 (Other: Johnson & Johnson Pharmaceutical Research & Development, L.L.C.); NCT01336504 (obsolete NCT alias)
Record Dates: First submitted 2002-12-09; First posted 2002-12-10 (Estimated); Last update posted 2013-01-10 (Estimated); Status verified 2013-01

CONDITIONS: Ovarian Neoplasms; Endocrine Gland Neoplasms; Neoplasms by Site; Neoplasms; Ovarian Diseases; Adnexal Diseases; Genital Diseases, Female
Keywords: Ovarian cancer; Ovary; Cancer; Trabectedin; Yondelis; ET743; Ecteinascidin 743; Antineoplastic Agents, Alkylating; Alkylating Agents
MeSH Terms: conditions — Ovarian Neoplasms; Endocrine Gland Neoplasms; Neoplasms by Site; Neoplasms; Ovarian Diseases; Adnexal Diseases; Genital Diseases, Female | interventions — Trabectedin; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Trabectedin (Experimental): Trabectedin 0.58 mg/m2 administered as a 3-hour intravenous infusion, Days 1, 8, and 15 every 28 days for up to approximately 3 years in the absence of disease progression. Dexamethasone 10 mg administered intravenously 30 minutes prior to each trabectedin infusion.
  Interventions: Drug: Trabectedin; Drug: Dexamethasone

INTERVENTIONS:
Drug: Trabectedin — Trabectedin 0.58 mg/m2, administered as a 3-hour intravenous infusion, Days 1, 8, and 15 every 28 days for up to approximately 3 years in the absence of disease progression.
Drug: Dexamethasone — Dexamethasone 10 mg administered intravenously 30 minutes prior to each trabectedin infusion.

SUMMARY:
The purpose of this study is to test the safety and effectiveness of an investigational chemotherapy agent in patients with advanced ovarian cancer.

DETAILED DESCRIPTION:
Patients will be enrolled in the study after all study-specific entry criteria are met and informed consent is obtained. Patients will be required to attend regular clinic visits to receive study medication and have their status monitored. Patients will also be required to have radiologic tumor assessments performed at multiple times throughout the study. A detailed explanation can be provided by the study physician (Investigator) conducting this study. Trabectedin at a starting dose of 0.58 mg/m2 will be given to patients intravenously (i.v). as a 3-hour infusion every week for 3 weeks (on Days 1, 8, and 15) of a 4 week cycle via a central venous catheter (also referred to as a "central line" which is a tube ie, "catheter" placed into a large vein). All patients will receive dexamethasone 10 mg i.v. 30 minutes prior to each trabectedin infusion. Patients may receive multiple cycles of trabectedin in the absence of disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of advanced epithelial ovarian cancer
* Progression or recurrence during or after platinum-containing regimen
* At least one measureable tumor lesion
* Adequate bone marrow, hepatic and renal function
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1

Exclusion Criteria:

* Known hypersensitivity to any components of the i.v. formulation of trabectedin or dexamethasone
* Pregnant or lactating women
* Known metastases (spread) of cancer to the central nervous system
* History of another neoplastic disease unless in remission for five years or more.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2002-10; Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Number of patients with objective response | Up to approximately 3 years

SECONDARY OUTCOMES:
The number of patients with an unbiased objective response | Up to approximately 3 years
Progression-free survival | Up to approximately 3 years
Time to progression | Up to approximately 3 years
Overall survival | Up to approximately 3 years
Duration of response | Up to approximately 3 years
Duration of stable disease | Up to approximately 3 years
Cancer antigen 125 (CA125) response | Up to approximately 3 years
The number of patients with adverse events | Up to approximately 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: Krasner CN, McMeekin DS, Chan S, et al. A Phase II study of trabectedin single agent in patients with recurrent ovarian cancer previously treated with platinum-based regimens. British Journal of Cancer. 2007:97:1618-24. — http://www.nature.com/doifinder/10.1038/sj.bjc.6604088